CLINICAL TRIAL: NCT00890812
Title: Factor XI Levels in Acute Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Sheila B. Terry Memorial Research Fund (Other)
Responsible Party: Jennifer Majersik, MD, University of Utah
Other Study IDs: 14363; ACC: 46499140; IRB: 00014363
Record Dates: First submitted 2009-04-28; First posted 2009-04-30 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Stroke
Keywords: Acute Ischemic Stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — A small 2ml vial of spun plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Factors VIII, IX and XI levels measured: Case group
- Non Stroke patients: This is the control group. This group represents patients who were initially evaluated for stroke.

SUMMARY:
The purpose of this study is to evaluate the utility of measuring coagulation factor activities in the setting of acute ischemic stroke, as potential markers of inherited thrombotic risk. The investigators will determine if relationships exist between coagulation factors, including factor VIII, factor IX, and factor XI and clinical diagnosis, classification, and outcome. The investigators will determine if any significant elevations of these factor activities are independent thrombotic risk factors.

Null Hypothesis: There is no statistical difference between coagulation factors, including factors VIII, IX, or XI activity levels in patients having acute ischemic stroke as compared to acute stroke mimics.

DETAILED DESCRIPTION:
Increased factor XI levels have been associated with venous thromboembolic disease and acute myocardial infarction. However, checking factor XI levels is not currently indicated to assess individual thromboembolic risk. Factor XI is an important protease that links the extrinsic arm of the coagulation cascade with the intrinsic arm through dual activation by both factor XII and thrombin. Since thrombin is a downstream product of factor XI, a feedback loop is created that amplifies thrombin production and ultimately results formation of a stable fibrin clot. Sufficient thrombin generation via this pathway also contributes to activation of the Thrombin-Activatable Fibrinolysis Inhibitor (TAFI). Activated TAFI downregulates fibrinolysis and has been implicated as part of the association between elevated factor XI levels and venous thromboembolic disease. One study found that functional TAFI levels of > 120% increased the risk of ischemic stroke approximately 6-fold, however, the association between Factor XI and ischemic stroke has yet to be firmly established. We recently performed a preliminary retrospective analysis of 78 patients with stroke or transient ischemic attack (TIA) and found that patients with factor XI activity levels above the 95th percentile of an age and sex matched reference population had a relative risk of 5.3 for stroke or TIA. Factor XI measurements may be able to help identify thromboembolic disease, aiding in the determination of stroke etiology.

ELIGIBILITY:
Inclusion Criteria:

* Those clinically diagnosed with acute ischemic stroke
* 18 years of age or greater

Exclusion Criteria:

* Those without clinical diagnosis of acute ischemic stroke will be included in the control group.
* Patients with hemorrhagic strokes
* Inpatients who are evaluated through the Brain Attack protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients presenting to the University of Utah Health Sciences Center Emergency Department.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2009-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To determine the relationship between elevated factors VIII, IX and XI and acute ischemic stroke as compared to other emergent events. | At time of incident stroke (baseline) and at early follow-up (30-60 Days post stroke).

SECONDARY OUTCOMES:
To determine the relationship between elevated factors VIII, IX and XI and stroke subtype. | 30-60 Days post stroke
To determine if a relationship exists between elevated factors VIII, IX and XI and the clinical severity and stroke outcome. | 30-60 Days post stroke
To determine if factors VIII, IX and XI level are different in the acute phase of ischemic stroke relative to chronic phase. | 30-60 Days post stroke
To determine if a relationship exists between factors VIII, IX and XI levels and early stroke/TIA recurrence. | 30-60 Days post stroke

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Majersik, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Health Sciences Center, Salt Lake City, Utah, United States

REFERENCES:
- [Result] Chandler WL, Rodgers GM, Sprouse JT, Thompson AR. Elevated hemostatic factor levels as potential risk factors for thrombosis. Arch Pathol Lab Med. 2002 Nov;126(11):1405-14. doi: 10.5858/2002-126-1405-EHFLAP. PMID 12421150
- [Result] Meijers JC, Tekelenburg WL, Bouma BN, Bertina RM, Rosendaal FR. High levels of coagulation factor XI as a risk factor for venous thrombosis. N Engl J Med. 2000 Mar 9;342(10):696-701. doi: 10.1056/NEJM200003093421004. PMID 10706899
- [Result] Minnema MC, Peters RJ, de Winter R, Lubbers YP, Barzegar S, Bauer KA, Rosenberg RD, Hack CE, ten Cate H. Activation of clotting factors XI and IX in patients with acute myocardial infarction. Arterioscler Thromb Vasc Biol. 2000 Nov;20(11):2489-93. doi: 10.1161/01.atv.20.11.2489. PMID 11073857
- [Result] Murakami T, Komiyama Y, Masuda M, Karakawa M, Iwasaka T, Takahashi H. Evaluation of factor XIa-alpha 1-antitrypsin in plasma, a contact phase-activated coagulation factor-inhibitor complex, in patients with coronary artery disease. Arterioscler Thromb Vasc Biol. 1995 Aug;15(8):1107-13. doi: 10.1161/01.atv.15.8.1107. PMID 7627703
- [Result] Santamaria A, Oliver A, Borrell M, Mateo J, Belvis R, Marti-Fabregas J, Ortin R, Tirado I, Souto JC, Fontcuberta J. Risk of ischemic stroke associated with functional thrombin-activatable fibrinolysis inhibitor plasma levels. Stroke. 2003 Oct;34(10):2387-91. doi: 10.1161/01.STR.0000088642.07691.15. Epub 2003 Aug 28. PMID 12947154
- [Result] Yang DT, Flanders MM, Kim H, Rodgers GM. Elevated factor XI activity levels are associated with an increased odds ratio for cerebrovascular events. Am J Clin Pathol. 2006 Sep;126(3):411-5. doi: 10.1309/QC259F09UNMKVP0R. PMID 16880142
- [Result] Salomon O, Steinberg DM, Koren-Morag N, Tanne D, Seligsohn U. Reduced incidence of ischemic stroke in patients with severe factor XI deficiency. Blood. 2008 Apr 15;111(8):4113-7. doi: 10.1182/blood-2007-10-120139. Epub 2008 Feb 11. PMID 18268095